CLINICAL TRIAL: NCT02450981
Title: Multicentre Open Label Non-randomized Clinical Study Evaluating Pharmacokinetics, Safety, Tolerability of Multiple Intravitreal Injections of BCD-021 (CJSC BIOCAD, Russia) in Patients With Neovascular Wet Age-related Macular Degeneration
Brief Title: Evaluation the Pharmacokinetics, Safety, Tolerability of BCD-021 in Patients With Neovascular Age-related Macular Degeneration
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BCD-021-1
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Neovascular Age-related Macular Degeneration
MeSH Terms: interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCD-021 group (Experimental): BCD-021 (bevacizumab) at a dose of 1.25 mg, administered as single intravitreal injection every 28 days up to 12 months.
  Interventions: Drug: Bevacizumab (BCD-021)

INTERVENTIONS:
Drug: Bevacizumab (BCD-021) — Bevacizumab is a monoclonal antibody against vascular endothelial growth factor A (VEGF-A)
  Other Names: Avastin

SUMMARY:
This clinical study is a phase 1 study which carried out to to evaluate the safety, pharmacokinetics and tolerability of multiple intravitreal injections of BCD-021(bevacizumab biosimilar candidate manufactured by CJSC BIOCAD, Russia) when used in patients with neovascular wet age-related macular degeneration.

DETAILED DESCRIPTION:
BCD-021-1 is an open label, non-comparative, non-randomized, multicenter phase 1 clinical study evaluating pharmacokinetics, safety and tolerability of multiple intravitreal injections of BCD-021 (bevacizumab biosimilar, CJSC BIOCAD) when given in patients with exudative (wet) age-related macular degeneration.

The study will enrol 10 patients with confirmed neovascular wet age-related macular degeneration. Before inclusion into the active phase of the study, patients will undergo a diagnostic examination during the screening period with a maximum duration of 28 days.

The principal part of the study includes the period from the first intravitreal injection and until 28 days after the third intravitreal injection. The goal of this stage is to evaluate pharmacokinetics, the safety and tolerability of multiple intravitreal injections of BCD-021 (CJSC BIOCAD, Russia) when used in patients with neovascular wet age-related macular degeneration.

Extension phase of the study (month 4 - month 12) is required to assess the long-term effects of the therapy and get full information about the immunogenicity of the study drug.

ELIGIBILITY:
Inclusion Criteria:

* subject has provided informed consent;
* men and women;
* patients must be from 50 years old;
* wet AMD in the study eye, defined as active choroidal neovascular membrane (CNV) (not previously treated with intravitreal injection of an anti-VEGF drug), including retinal angiomatous proliferation (RAP), with oedema involving the fovea as demonstrated with optical coherence tomography (OCT);
* best corrected VA for the studied eye ranging between 20/32 (6.3/10) and 20/320 (0.6/10) with ETDRS scale;
* size of lesion < 12 disk area;
* in case of occult neovessels, proof required of recent development of the lesion: loss of VA of at least 5 letters ETDRS in the last 3 months OR appearance of a subretinal hemorrhage OR increase in the size of the lesion (> 10%) using fluorescein angiography during the last month by comparison with the last 3 months OR appearance of OCT criteria of macular oedema type, serous separation of neuro-epithelium, separation of the pigmented epithelial during the last month before inclusion to trial;
* only one eye of each study patient may be recruited into the study;
* patient's ability to follow the protocol procedures;
* male and female patients with normal reproductive function and their sexual partners are aware and willing to use voluntarily reliable methods of contraception during the whole period of the study including the screening period.

Exclusion Criteria:

* Previous or current treatment with intravitreal injection of an anti-VEGF drug (ranibizumab, bevacizumab, aflibercept or pegaptanib, etc.);
* Other healing treatment in the studied eye during the last 3 months before the first injection;
* Former vitrectomy in the study eye;
* Medical history of photocoagulation in the studied eye;
* Involvement in another clinical study (studied eye and/or the other eye);
* Subretinal hemorrhage reaching the fovea centre, with a size > 50% of the lesion area;
* Fibrosis or retrofoveal retinal atrophy in the studied eye;
* Retinal pigment epithelial tear reaching the macula in the studied eye;
* Choroidal neovascularisation not related to a AMD in the studied eye;
* Medical history of intravitreal medical device in the studied eye;
* Active or suspected ocular or peri-ocular infection;
* Acute conjunctivitis, keratitis, scleritis, or endophthalmitis;
* Serious active intra-ocular inflammation in the studied eye;
* Macula-foramen of the studied eye;
* Myopia larger than -8 diopter;
* Former corneal grafting of the studied eye;
* Medical history of auto-immune or idiopathic uveitis;
* Proved diabetic retinopathy;
* Intra-ocular pressure ≥ 25 mmHg despite two topical hypotonic treatments;
* Medical history of intra-ocular surgery within 2 months before the first injection in the studied eye;
* Aphakia or lack of lens capsule (not removed by laser) in the studied eye;
* Any illness or ocular condition that would require an intra-ocular surgery in the studied eye within 12 months after the inclusion;
* Known hypersensitivity to bevacizumab or another drug composite of the medicinal products used; allergy to anaesthetic eye drops;
* Arterial hypertension that is not controlled by an appropriate treatment;
* Previous or current treatment with systemic administration of bevacizumab;
* Pregnancy and breast-feeding;
* Any determined immunodeficiency;
* Syphilis, HIV, hepatitis B, any history of hepatitis C virus;
* Any mental disorder that can create a risk for the patient or influence the patient's ability to follow the study protocol;
* Drug addiction, alcoholism.
* Presence or history of malignant neoplasm (including lymphoproliferative disease);
* Simultaneous participation in any other clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Frequency of ocular and systemic AEs (adverse events) and SAEs (serious adverse events) which are related to BCD-021 and appeared after the first, the second and the third intravitreal injection of BCD-021 | 85 days

SECONDARY OUTCOMES:
Frequency of ocular and systemic AEs and SAEs related to age-related macular degeneration (AMD) therapy, appeared within the whole study period | 12 months
Number of cases of early withdrawal from the study caused by AE or SAE | 12 months
Area under the plasma concentration-time curve from zero (0) hours to 28 days, maximum concentration and half life of bevacizumab after the first administration of BCD-021 | 28 days
Area under the plasma concentration-time curve from 56 days to 84 days, maximum concentration and half life of bevacizumab after the third administration of BCD-021 | 28 days
Minimum concentration of bevacizumab between the first and the third administration of BCD-021 | 28 days
Number of patients who have binding and neutralizing antibodies to BCD-021 in serum at screening, after 3 intravitreal injections and after 12 intravitreal injections of BCD-021 | 12 months
Mean change in visual acuity score, measured on the Early Treatment Diabetic Retinopathy Study (ETDRS) scale at month 12 | 12 months
Change in fluid and foveal thickness on OCT during the study | 12 months
Timing of visual improvement after initiation of therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, Phd, Study Chair — CJCS BIOCAD